CLINICAL TRIAL: NCT05747287
Title: A Post-Market Study to Evaluate the Safety and Efficacy of Pronavi Microcatheter for Use in Endovascular Interventions
Brief Title: Evaluate Safety and Efficacy of Pronavi Microcatheter for Use in Endovascular Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BrosMed Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S02
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Peripheral Arterial Disease
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Device: microcatheter

INTERVENTIONS:
Device: microcatheter — supports the insertion of the guide wire，exchange of the guide wire and the delivery of contrast media

SUMMARY:
This is a prospective, multi-center, single-group post-market study. It is planned to be carried out in about 3 clinical institutions, and a total of 60 subjects are expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Patients with symptomatic ischemic heart disease who are suitable for non-acute percutaneous coronary intervention (PCI);
3. Patients with target lesion diameter stenosis ≥ 70% (visually) or de novo coronary chronic total occlusion (CTO), or tortuous lesions, who plan to use Pronavi Microcatheter;
4. Patients or their guardians who understand the purpose of the trial, voluntarily participate and sign the written informed consent, and are able to be followed up.

Exclusion Criteria:

1. Patients with clinical symptoms consistent with ST-elevation myocardial infarction and/or ECG changes within 12 hours before the procedure;
2. Patients who are known to be intolerant to antiplatelet drugs or allergic to contrast media;
3. Patients with in-stent occlusion;
4. Patients with unprotected left main coronary artery disease;
5. Women who are pregnant or lactating;
6. Patients who are participating in clinical trials of other drugs or medical devices;
7. Patients with contraindications to the investigational device;
8. Other patients considered by the investigators to be unsuitable for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Technical success | 0 day
  Defined as successful guide wire passage, that is, the Pronavi Microcatheter successfully supports the guide wire through the target lesion to reach the distal true coelom.

SECONDARY OUTCOMES:
Device success | 0 day
  Defined as delivery of the microcatheter to the designated site, assistence of guide wire into the target vessel, and successful withdrawal.
Procedural success | 0 - 7 days
  Defined as meeting all the following criteria:
  1. After PCI, the final diameter stenosis of the target lesion achieves ≤30%, and the TIMI returns to grade 3;
  2. No all-cause death, Q-wave myocardial infarction, stroke, cardiac tamponade, target vessel revascularization (including re-PCI or emergency coronary artery bypass grafting) before discharge.
Device super-selective angiography (if applicable) | 0 day
  the microcatheter shall deliver the contrast agent to the designated location and develop
Guide wire exchange supported (if applicable) | 0 day
  successful exchange of the guide wire
Device Performance Evaluation | 0 day
  The investigators will evaluate the device performance according to the use and operation of the device during the procedure

OTHER OUTCOMES:
Major adverse cardiac events (MACE) during the study | 0 - 7 days
  Major adverse cardiac events (MACE) are defined as cardiac death, myocardial infarction, and target lesion revascularization (TLR).
Adverse events and serious adverse events related to the study device during the study | 0 - 7 days
Occurrence of other adverse events and serious adverse events during the study | 0 - 7 days

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - The Seventh People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No